CLINICAL TRIAL: NCT03065621
Title: Neoadjuvant Biomarker ResearcH Study of Palbociclib Combined With Endocrine Therapy in Estrogen Receptor Positive/HER2 Negative Breast CAncer
Brief Title: Neoadjuvant Biomarker ResearcH Study of Palbociclib Combined With Endocrine Therapy in Estrogen Receptor Positive/HER2 Negative Breast CAncer (NeoRHEA)
Acronym: NeoRHEA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IJB-BC-NEORHEA-2016
Record Dates: First submitted 2017-01-12; First posted 2017-02-28 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2020-08

CONDITIONS: Breast Cancer Female
Keywords: Breast
MeSH Terms: interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Palbociclib with Endocrine Therapy (Experimental): All subjects will receive palbociclib 125 mg for 4 cycles, orally, once a day, for 21 days followed by 7 days of rest (4 cycles of 28 day long). After the final rest week (therefore post cycle 4), subjects will receive 3 to 7 additional days of palbociclib, as necessary, at the same dose and posology, until the day before curative intent surgery. Depending upon the menopausal status, the patient will receive either letrozole or tamoxifen continuously during the palbociclib treatment (which consists of 4 cycles of 28 days).
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Each cycle will be 28 days. Patient will take study drug daily during 21 days and then have a rest period of 7 days.
  Other Names: PD-0332991; Ibrance

SUMMARY:
This is an open-label, single arm, phase 2 trial that will include pre or post-menopausal female subjects, that have ER-positive, HER2-negative early breast cancer. Subject will receive 4 cycles of palbociclib 125 mg (each cycle of palbociclib consists of treatment from D1 to D21 followed by a week of rest) combined with endocrine therapy given continuously (each cycle of endocrine therapy consists of treatment from D1 to D28).

The endocrine therapy will be determined according to the menopausal status of the subject evaluated at the study screening.

DETAILED DESCRIPTION:
This is an open-label, single arm, phase 2 trial that will include pre or post-menopausal female subjects, that have ER-positive, HER2-negative early breast cancer. Subject will receive 4 cycles of palbociclib 125 mg (each cycle of palbociclib consists of treatment from D1 to D21 followed by a week of rest) combined with endocrine therapy given continuously (each cycle of endocrine therapy consists of treatment from D1 to D28).

The endocrine therapy will be determined according to the menopausal status of the subject evaluated at the study screening.

For post-menopausal subjects: endocrine therapy will consist of letrozole 2.5 mg continuously.

For pre-menopausal or peri-menopausal subjects: endocrine therapy will consist of tamoxifen 20 mg continuously, combined or not with goserelin 3.6 mg monthly at the local investigator's discretion.

Endocrine therapy for both groups should continue until the last day of palbociclib treatment (i.e. the day before surgery).

Subject's response to therapy will be evaluated before and after the 4 cycles of treatment by ultrasound to determine response to therapy. Post treatment ultrasound should be performed 7 to 10 days before surgery (with a maximum delay of 3 days in case of delayed surgery date).

Surgery will be performed 4 to 8 days after the end of the 4th cycle of study treatment.

Biopsy samples will be collected after the subject's inclusion in the study and prior to Day 1 Cycle 1 of study treatment (pre-treatment biopsy) and will consist of collection of 4 core biopsies (2 FFPE and 2 Frozen).

FFPE and frozen material will be collected from the surgical material left over, after sufficient and relevant parts has been retained to establish, improve or complement the diagnosis or treatment of the subject.

One whole blood sample (1x10 mL) will also be collected after the subject's inclusion and prior to Day 1 Cycle 1 of study treatment.

Blood samples for plasma processing (4x10 mL per time point) will be collected after the subject's inclusion and prior to Day 1 Cycle 1, prior to Day 1 Cycle 2 of study treatment, at surgery day (prior surgery) and one month after surgery.

All the biological samples collected (pre-treatment biopsy, material from surgery and all blood samples) within the study are mandatory. The breast biopsy samples as well as imaging tumour assessment (ultrasound breast) performed prior to the signature of the study ICF are not admissible for assessment of study end-points and should be repeated within the required study time window.

Information on patient survival and disease recurrence will be collected at least 30 months from the date of the end of study treatment (i.e., last visit of the last subject one month after surgery day, see definition in paragraph 11.3). Data collection will be made based on medical charts if a follow up visit was performed not earlier than February 2022. If the data is missing from medical charts (i.e. loss of follow up), a phone call to the subject's general practitionerwill be made.

Primary objective :

• To identify biomarkers of resistance to a 4-month preoperative treatment of palbociclib plus endocrine therapy defined as stable or progressive disease by ultrasound (based on WHO criteria) using RNA-seq of the baseline tumour biopsy.

Secondary objectives :

* To identify biomarkers of resistance to a 4-month preoperative treatment of endocrine therapy and palbociclib by correlating tumour response by ultrasound (mandatory) or magnetic resonance (optional) imaging (response will be assessed as continuous or categorical variable) with RNA-seq of the baseline tumour biopsy
* To identify biomarkers of resistance to a 4-month preoperative treatment of palbociclib plus endocrine therapy defined as residual disease burden, RCB of 3 using RNA-seq of the baseline tumour biopsy
* To identify biomarkers of resistance to a 4-month preoperative treatment of endocrine therapy and palbociclib defined as GGI high by RNA-seq of the residual tumour at surgery using RNA-seq of the baseline tumour biopsy
* To understand mechanisms of resistance to the combination of endocrine therapy and palbociclib by comparing the transcriptome of tumours at baseline and at surgery using RNA-seq
* To evaluate the safety of the combination of palbociclib plus endocrine therapy
* To evaluate the role of plasma ctDNA in monitoring response/resistance to pre-operative treatment with endocrine therapy and palbociclib
* To validate/further refine an 11-gene expression signature associated with response/resistance to palbociclib and endocrine treatment

Exploratory objectives:

* To compare changes in clonal composition, transcriptomic changes and changes in the open chromatin state of tumour cells using a combined genomic and transcriptomic (G&T) single tumour cell analysis and chromatin accessibility single tumour cell analysis of exceptional responders and exceptional non-responders. Based on the above results, additional bulk or single cell analyses in the entire study cohort could be performed.
* To evaluate associations between patient survival (distant relapse-free survival, relapse-free survival, invasive disease-free survival, overall survival) and the following :

  * Tumor clinicopathological characteristics and other biomarkers at baseline and/or surgery and/or their changes
  * Plasma ctDNA monitoring

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age ≥ 18 years
3. Histological diagnosis of breast adenocarcinoma that is estrogen receptor-positive, and HER2- negative as per the updated American Society of Clinical Oncology (ASCO) - College of American Pathologists (CAP) guidelines according to local testing.
4. Multifocal unilateral or bilateral breast adenocarcinoma tumours are allowed provided that all tested foci are ER-positive and HER2-negative.

   * ER-positive (ER+ is defined as having a IHC of 1% or more and/or and Allred of 2 or more and HER2-negative.
   * HER2 negative (HER2 negative is defined as having an IHC of 1+ without ISH OR IHC 2+ and ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells OR ISH non-amplified with ratio less than 2.0 and if reported, average HER2 copy number < 4 signals/cells (without IHC)
5. A primary non metastatic or locally advanced tumour of more than 2 cm (T2 or T3), N0 or N1 without prior treatment candidate for preoperative treatment
6. ECOG Performance Status (PS) 0 or 1.
7. Adequate Bone Marrow Function including:

   1. Absolute Neutrophil Count (ANC) ≥1500/μL or ≥1.5 x109/L;
   2. Platelets ≥100000/μL or ≥100 x 109/L;
   3. Hemoglobin ≥ 9 g/dL.
8. Adequate Renal Function including: Serum creatinine ≤ 1.5 x upper limit of normal (ULN) or estimated creatinine clearance ≥ 60 ml/min as calculated using the method standard for the institution.
9. Adequate Liver Function, including all of the following parameters:

   1. Total serum bilirubin ≤ 1.0 x ULN unless the subject has documented Gilbert syndrome (in which case up to 3 x ULN is acceptable) ;
   2. Aspartate and Alanine Aminotransferase (AST and ALT) ≤ 1.5 x ULN;
   3. Alkaline phosphatase ≤ 2.5 x ULN.
10. Signed consent form
11. Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests, radiological exams, tumour and blood specimen collection and other procedures.
12. Women who are not postmenopausal or have not undergone hysterectomy must have documented negative pregnancy test (serum) prior to inclusion.
13. Female subjects of child bearing potential and their partners, who are sexually active, must agree to the use of two highly effective forms of contraception in combination throughout the period of taking study treatment and for at least 90 days after last dose of study drug, or they must totally/truly abstain from any form of sexual intercourse. Use of oral hormonal contraceptive agents in this study is not permitted.

Exclusion Criteria:

1. Clinical T4 disease including inflammatory breast cancer.
2. Prior history of invasive cancer including breast cancer except basal or squamous cell carcinoma of skin that has been definitively treated.
3. Known hypersensitivity to the study drugs or excipients.
4. Any illness or medical condition that is unstable or could jeopardize the safety of the subject or her compliance with study requirements.
5. Subjects unable to swallow oral medications.
6. Prior intake of letrozole, or any CDK inhibitor or anti-cancer therapy.
7. Concurrent treatment with any of the drugs not permitted, i.e. strong CYP3A inhibitors/inducers and drugs known to cause QTc interval prolongation (see section 5.7 for specific instructions).
8. QTc exceeding 480 msec, family or personal history of long or short QT syndrome, Brugada syndrome or known history of QTc prolongation, or Torsade de Pointes (TdP).
9. Uncontrolled diabetes, according to investigator's clinical judgment.
10. Pregnant or lactating women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
To identify biomarkers of resistance to a 4-month preoperative treatment of palbociclib plus endocrine therapy defined as stable or progressive disease by ultrasound (based on WHO criteria) using RNA-seq of the baseline tumour biopsy | 4 Months
  • Baseline transcriptomic profile of resistance to 4 months of palbociclib and endocrine therapy defined as stable or progressive disease by ultrasound based on WHO criteria

SECONDARY OUTCOMES:
To identify biomarkers of resistance to a 4-month preoperative treatment of endocrine therapy and palbociclib by correlating tumour response by ultrasound (mandatory) or magnetic resonance (optional) imaging | 4 Months
  • Baseline transcriptomic profile of resistance to 4 months of palbociclib and endocrine therapy assessed by ultrasound (mandatory) or magnetic resonance (optional) imaging (response will be assessed as continuous or categorical variable)
To identify biomarkers of resistance to a 4-month preoperative treatment of palbociclib plus endocrine therapy defined as residual disease burden, RCB of 3 using RNA-seq of the baseline tumour biopsy | 4 Months
  • Baseline transcriptomic profile of resistance to 4 months of palbociclib and endocrine therapy, defined as an RCB of 3.
To identify biomarkers of resistance to a 4-month preoperative treatment of endocrine therapy and palbociclib defined as GGI high by RNA-seq of the residual tumour at surgery using RNA-seq of the baseline tumour biopsy | 4 Months
  • Baseline transcriptomic profile of resistance to 4 months of palbociclib and endocrine therapy, defined as an GGI high at surgery
To understand mechanisms of resistance to the combination of endocrine therapy and palbociclib by comparing the transcriptome of tumours at baseline and at surgery using RNA-seq | 4 Months
  • Transcriptomic changes between pre-treatment and post-treatment tumour samples
To evaluate the safety of the combination of palbociclib plus endocrine therapy as assessed by the NCI-CTCAE version 4.03 | 4 Months
  Safety
The role of plasma ctDNA in monitoring response/resistance to pre-operative treatment with endocrine therapy and palbociclib | 4 Months
  • Plasma ctDNA analysis to monitor response/resistance to pre-operative treatment with endocrine therapy and palbociclib
To refine an 11-gene expression signature associated with response/resistance to palbociclib and endocrine treatment | 4 Months
  • Validation of 11-gene expression signature associated with response/resistance to palbociclib and endocrine treatment
To determine the effect of a pre-operative treatment with endocrine therapy and palbociclib on anti-tumour immune response | 4 Months
  • Changes in anti-tumour immune response between pre- and post-treatment tumour samples
To determine the effect of a pre-operative treatment with endocrine therapy and palbociclib on tumour senescence | 4 Months
  • Changes in tumour senescence between pre- and post-treatment tumour samples

OTHER OUTCOMES:
To compare changes in clonal composition, transcriptomic changes and changes in the open chromatin state of tumour cells | 4 Months
  chromatin accessibility single tumour cell analysis of exceptional responders and exceptional non-responders
To compare changes in clonal composition, transcriptomic changes and changes in the open chromatin state of tumour cells | 4 Months
  combined genomic and transcriptomic (G&T) single tumour cell analysis
Distant relapse-free survival (DRFS) | 36 months
  time between breast surgery and the date of diagnosis of distant recurrence or death from any cause
Relapse-free survival (RFS) | 36 months
  time between breast surgery and the date of diagnosis of distant or locoregional invasive recurrence or death from any cause
Invasive disease-free survival (iDFS) | 36 months
  time between breast surgery and the date of diagnosis of local or distant invasive recurrence
Overall survival (OS) | 36 months
  time between surgery and the day of death (due to any causes) or day of last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michail Ignatiadis, MD, Study Chair — Jules Bordet Institute
Locations (5):
- Belgium (5):
  - Institut Jules Bordet, Anderlecht
  - CHU Brugmann, Brussels
  - CHU Saint-Luc, Brussels
  - UZ Leuven Gasthuisberg, Leuven
  - CHU UCL Namur Sainte-Elisabeth, Namur

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papagiannis A, Majjaj S, Duhoux FP, Agostinetto E, Stanciu AM, Vanhulst T, Buisseret L, Larsimont D, Veys I, Paesmans M, Hammer TB, Awada A, Ameye L, Rothe F, Madriles F, Cash TP, Salgado R, Willard-Gallo K, Sotiriou C, Vuylsteke P, Neven P, Ignatiadis M. Palbociclib and endocrine therapy diminish adaptive anti-tumor immunity in early breast cancer: The NeoRHEA phase 2 study. Nat Commun. 2025 Nov 26;16(1):11659. doi: 10.1038/s41467-025-66590-2. PMID 41298425
- [Derived] Brandao M, Coens C, Ignatiadis M. Patient-reported outcomes and genomic signatures: tools to tailor adjuvant endocrine treatment? Ann Oncol. 2019 Nov 1;30(11):1677-1681. doi: 10.1093/annonc/mdz404. No abstract available. PMID 31613310